Statistical Analysis plan

Version 1: 21.07.2025

Title: A secondary analysis of the PEACH study data to investigate the impact of a penicillin allergy record on antibiotic use, AMR and patient health outcomes in patients admitted with COVID-19

1 Introduction

1.1 BACKGROUND AND RATIONALE

Coronavirus disease (COVID-19) is a viral respiratory tract infection caused by the SARS-CoV-2 virus. Antibiotics are often used in patients with COVID-19 because: a) there is clinical difficulty in distinguishing bacterial pneumonia from COVID-19 or b) there are concerns about co-infection either at the time of presentation or as a secondary infection related to COVID-19 or hospital admission. A large meta-analysis which included 30,623 patients, found that 74.6% (95% CI 68.3-80.0%) of inpatients with COVID-19 were prescribed antibiotics. Despite the antibiotic usage in this cohort, systematic reviews have found the prevalence of bacterial infections to be only 7-9%, highlighting that antibiotic prescribing in this cohort is often inappropriate.<sup>2-4</sup>

The impacts of PenA on antibiotic prescribing and AMR in patients with COVID-19 is largely unknown. One United States based retrospective study investigating the impact of PenA on outcomes for patients with COVID-19 found that rates of hospitalisation, intensive care admission, acute respiratory failure, and mechanical ventilation were higher in patients with PenA compared to those without PenA.<sup>5</sup> This risk remained even in the absence of bacterial infection. Studies exploring this further are required. However, if we extrapolate from pre-pandemic data, we can hypothesise that patients hospitalised with COVID-19 with PenA and treated for bacterial infections, will be at risk of longer hospital stays, higher rates of treatment failure and have higher mortality when compared to patients without PenA.

This analysis will explore the impact of PenA on outcomes for patients COVID-19 in the UK, by conducting a secondary analysis of data from the PEACH (Procalcitonin: Evaluation of Antibiotic use in COVID-19 Hospitalised patients) study.

PEACH was a retrospective cohort study aimed at determining if the use of a biomarker for infection called procalcitonin (PCT) reduced antibiotic use among patients who were hospitalised with COVID-19 during the first wave of the pandemic. As such this data set will have data pertaining to antibiotic use, allergy status, AMR and patient outcomes that will allow investigation of the impact PenA has on this patient group.

#### 1.2 STUDY OBJECTIVES AND HYPOTHESIS

The study objective is to examine the relationship between PenA labels and AMR and patient health outcomes in patients admitted with COVID-19. Our hypothesis is that patients with penA will be higher rates of adverse health outcomes such as death and AMR infections.

## 2 STUDY METHODS

#### 2.1 STUDY DESIGN AND DATA SOURCE

Secondary analysis of PEACH study data. The PEACH study was a multi-centre, retrospective, observational, cohort study using patient-level clinical data (IRAS: 290358) which investigated whether the use of procalcitonin testing, to guide antibiotic prescribing, safely reduced antibiotic use amongst hospitalised patients with COVID-19 during the first wave of the pandemic using routinely collected patient institutional clinical databases and patient medical records.<sup>6</sup> Data were collected in 11 NHS acute hospital Trusts and Health Boards in England and Wales, and data in a pseudo-anonymised format was received from the Cardiff Clinical Trials Unit who were the data controllers for the PEACH study. This study has been designed in accordance with the STROBE (Strengthening the Reporting of Observational Studies in Epidemiology) guidelines, which will also be followed in the reporting of results.<sup>7</sup>

## 2.2 SAMPLE SIZE CALCULATION

Mortality in COVID-19 patients in the first wave of the pandemic was approximately 30%. Therefore using 5% significance level, a sample size of 7000 will provide 80% statistical power to detect a change of 4.5% or greater in mortality.

### 2.3 TIMING OF FINAL ANALYSIS

Analysis will be conducted once data has been received by the PEACH study team.

# 3 STATISTICAL PRINCIPLES

### 3.1 CONFIDENCE INTERVALS AND P-VALUES

All hypothesis tests and confidence intervals will be two-sided. A significance level of 0.05 will be used, and results will be presented with 95% confidence intervals.

### 3.2 ANALYSIS POPULATION

PEACH study participants which includes patients ≥16 years admitted to a participating NHS hospital and diagnosed with COVID-19 between 01/02/2020 and 30/06/2020. Only participants with their penicillin allergy status recorded will be included in the analysis population.

## 4 STUDY POPULATION

## 4.1 POPULATION

#### 4.1.1 Inclusion criteria

Adult (>16 years) with confirmed COVID-19 (positive PCR test) and admitted to participating NHS Trusts/hospitals (for any reason) between 01/02/2020 to 30/06/2020.

#### 4.1.2 Exclusion criteria

Patients with their allergy status missing from the database will be excluded.

#### 4.2 BASELINE CHARACTERISTICS

Baseline data will include:

- Age
- Sex
- IMD
- Ethnicity
- Admission hospital
- Illness severity
- Co-morbidities

Baseline data were collected in the following sequence depending on availability: 1. Values on the day of COVID-19 test; 2. Values on day after COVID-19 test (if values on day of test are missing); and 3. Values on day before COVID-19 test (if values on day of test and values on day after the test are missing).

## 4.3 POTENTIAL CONFOUNDING COVARIATES

Directed Acyclic Graphs (DAG) display assumptions surrounding the exposure and outcome and serves as a tool to identify cofounder and mediators (which are responsible for part of the effect of the exposure). A DAG (Figure 1) was created a-priori to identify potential confounding variables that might affect both the exposure and outcome relating to AMR, this was developed based on existing literature and expert consensus within the supervisory team. Co-morbidities include: Asthma, cancer, CHD, CKD, COPD, diabetes, PAD, smoking, stroke and TIA.



Figure 1. Directed acyclic graph of the proposed associated between penA and AMR mediated by antibiotic exposure

## 4.4 PECO SUMMARY

| Population | Inpatients ≥16 years admitted with confirmed COVID-19 during hospital |
|---|---|
| | admission between 1 February 2020 and 30 June 2020. |
| Exposure | Presence of penicillin allergy record for the patient |
| Comparator | Patients without a penicillin allergy record |
| Outcomes | Primary: 60 day mortality |
| | Secondary outcomes: |
| | Presence antimicrobial resistant secondary bacterial infection |
| | Length of hospital stay |
| | Antibiotic usage in hospital |
| | Clostridioides difficile infection |
| | Treatment failure |
| | Day 30 mortality |

## 5 ANALYSIS

## 5.1 OUTCOME DEFINITIONS

### 5.1.1 Primary outcome

The primary outcome is mortality within 60 days of COVID-19 diagnosis in patients with and without a penA. This will be measured from the date of positive COVID 19 test.

## 5.1.2 Secondary outcomes

## 5.1.2.1 Presence antimicrobial resistant secondary bacterial infection

This will be determined by blood cultures and deep respiratory culture positivity. Blood culture results will are considered to be defined as the detection of bacteria according to Appendix, table 1 in a blood culture. A bacteraemia caused by potential skin contaminants (e.g. coagulase-negative staphylococci

[CoNS], *Corynebacterium* species, Bacillus species, *Cutibacterium* species, and *Micrococcus* species) will be considered to be significant if isolated in two or more blood cultures within a 48 hour period.<sup>10-12</sup> Deep respiratory cultures are considered to be positive if they grow a recognised pathogen as per the PEACH study protocol.

For the purpose of this study, the Magiorakos et al  $^{13}$  definition of resistance will be used and a infection will be considered to be a resistant infection if the isolated pathogen is resistant to  $\geq 1$  antibiotic agent in 3 or more antibiotic classes (Appendix, Table 2), antibiotic classes were derived from the WHO ATC/DDD Index 2024<sup>14</sup> and Mandel et al<sup>15</sup>.

#### 5.1.2.2 Length of hospital stay

Total hospital stay (day 0 = date of admission), calculated as days from admission date to the date of discharge or inpatient death (whichever occurred first).

#### 5.1.2.3 Antibiotic usage

Inpatient antibiotic use including antibiotic agent, route of administration and duration following COVID-19 diagnosis in hospital from day 1 of COVID-19 diagnosis to date of discharge or death (inclusive of day 1 and last day).

#### 5.1.2.4 Clostridioides difficile infection

As determined by a toxin positive result from day 1 of COVID-19 diagnosis

#### 5.1.2.5 Treatment failure

This will be defined as re-prescription of an antibiotic within 30 days of index antibiotic prescription

#### 5.1.2.6 Day 30 mortality

This will be measured from the date of positive COVID 19 test.

### 5.2 ANALYSIS METHODS

#### 5.2.1 Descriptive statistics

Descriptive statistics will be used to summarise baseline characteristics (Table 2) and types of antibiotics used stratified by exposure (penA status). Categorical data will be reported as percentages and frequencies and continuous data reported as medians with interquartile ranges (IQR) or as means with standard deviations (SD) depending on the distribution and characteristics of the data.

The chi-square test of association or the Fisher exact test will be used to test for relationships between categorical variables and the exposure. For continuous data, the Mann-Whitney U Test will be used for data that is not normally distributed and the independent t-test will be used for normally distributed data.

## Summary of baseline characteristics:

| | | | | Total | PenA | Non-PenA | p-value |
|-----|-----------|-------------|-------|-------|------|----------|---------|
| SD | D) or me | dian or IQI | R) | | | | |
| k | British, | Caribbea | an or | | | | |
| an | n British | | | | | | |
| ult | tiple eth | nic groups | | | | | |
| thr | nic grou | р | | | | | |
| mo | orbiditie | !S | | | | | |
| dit | ities | | | | | | |
| orb | bidity | | | | | | |
| om | morbiditi | es | | | | | |
| om | norbiaiti | es | | | | | |

| Γ | T | T | T |
|--------------------------------------------|---|---|---|
| Cancer, (n,%) | | | |
| Coronary heart disease, (n,%) | | | |
| CKD, (n,%) | | | |
| CVS, (n,%) | | | |
| Dementia, (n,%) | | | |
| Depression, (n,%) | | | |
| Epilepsy, (n,%) | | | |
| Heart Failure, (n,%) | | | |
| HTN, (n,%) | | | |
| Learning disability (LD), (n,%) | | | |
| Mental Health, (n,%) | | | |
| Obesity (BMI), (n,%) | | | |
| Osteoporosis, (n,%) | | | |
| PVD, (n,%) | | | |
| Palliative care, (n,%) | | | |
| RA, (n,%) | | | |
| Stroke (not transient), (n,%) | | | |
| Stroke (transient), (n,%) | | | |
| Liver disease (mild to severe), (n,%) | | | |
| HIV, (n,%) | | | |
| CTD, (n,%) | | | |
| Chronic neurological condition, (n,%) | | | |
| Smoker, (n,%) | | | |
| Primary care frailty score, mean (SD) or | | | |
| median or IQR) | | | |
| Admission site (n, %) | | | |
| Leeds | | | |
| Royal Liverpool | | | |
| Aneurin Bevan UHB | | | |
| Sheffield | | | |
| Cornwall | | | |
| Mid Yorkshire | | | |
| Bristol | | | |
| Brighton | | | |
| Newcastle | | | |
| Salford | | | |
| Nottingham | | | |
| COVID severity at time of diagnosis | | | |
| Baseline temperature, mean (SD) or median | | | |
| or IQR) | | | |
| qSOFA, mean (SD) or median or IQR) | | | |
| 4C mortality score, mean (SD) or median or | | | |
| IQR) | | | |
| Covid treatment Y or N | | | |
| Baseline CRP, mean (SD) or median or IQR) | | | |
| <u> </u> | | • | • |

| Baseline WCC, mean (SD) or median or IQR) |
|-------------------------------------------|
| ICU admission at diagnosis |

Descriptive statistics will also be used to summarise the antibiotic use (class of antibiotics, administration routes and duration of antibiotic use) within each exposure group.

#### 5.2.2 Explanatory analysis

For the primary and binary secondary outcome analysis, associations between exposure, covariates and outcome will be tested using multivariable logistic regression for binary outcomes. Multivariable regression will be reported as odds ratios (ORs) with 95% confidence intervals (CIs) and p-values.

For the two time to event outcomes (length of hospital stay and total days on antibiotics) a competing risks survival analysis will be undertaken to account for the possibility that some patients may die before these outcomes can be fully observed. Inpatient death will be treated as a competing event, and a cause-specific Cox proportional hazards model will be used, with results reported as hazard ratios (HRs) along with 95% confidence intervals (CIs) and p-values.

Confounders included in the regression analyses will include those identified a-priori from the DAG.

| | PenA (n/%) | Non PenA (n/%) | unadjusted<br>OR/HR (95%<br>CI) | adjusted<br>OR/HR<br>(95% CI) |
|---|---|---|---|---|
| Primary outcome | | | | |
| 60 day mortality | | | | |
| Secondary outcomes | | | | |
| Presence antimicrobial resistant secondary bacterial infection | | | | |
| Length of hospital stay | | | | |
| Total days antibiotic | | | | |
| Clostridioides difficile infection | | | | |
| Treatment failure | | | | |
| Day 30 mortality | | | | |

A sensitivity analysis will be conducted using a competing risks model for the remaining secondary outcomes to assess the potential impact of inpatient death as a competing event.

### 5.2.3 Missing data

Data may or may not be missing at random, therefore patterns of missingness will be explored and summarised descriptively by penA status.

The frequency (percentage) of missing data will be reported for baseline characteristics and for the study outcomes. Characteristics of those with and without missing values will be to explore reasons for missingness and whether data may be missing at random.

Subsequent to initial analyses, and where deemed appropriate, sensitivity analyses will be undertaken. For variables exhibiting more than 10% missing data, multiple imputation methods will be considered. Additionally, a sensitivity analysis incorporating a 'missing' category will be performed and compared against complete case analyses to assess the robustness of the findings.

## 5.2.4 Additional analysis

n/a

#### 5.2.5 Statistical software

Data will be analysed using R Studio, R version 4.3.3

# 6 APPENDIX

Appendix table 1. Categorisation of bacteria

| 0 /0: 10 | | |
|---|---|---|
| Genus/Clinical Group | Subgroup Classification | Organism |
| Staphylococcus aureus | Staphylococcus aureus | Staphylococcus aureus |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus capitis |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus caprae |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus cohnii |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus epidermidis |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus haemolyticus |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus hominis |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus saccharolyticus |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus saprophyticus |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus sciuri |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus spp. |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus warneri |
| Coagulase-negative Staphylococcus | Coagulase-negative Staphylococcus | Staphylococcus xylosus |
| Coagulase-negative Staphylococcus | Staphylococcus lugdunensis | Staphylococcus lugdunensis |
| Beta-haemolytic Streptococci | Group A Streptococcus | Streptococcus pyogenes |
| Beta-haemolytic Streptococci | Other beta haemolytic Streptococcus | beta Haemolytic Strep, group B |
| Beta-haemolytic Streptococci | Other beta haemolytic Streptococcus | beta Haemolytic Strep, group C |
| Beta-haemolytic Streptococci | Other beta haemolytic Streptococcus | beta Haemolytic Strep, group D |
| Beta-haemolytic Streptococci | Other beta haemolytic Streptococcus | beta Haemolytic Strep, group F |
| Beta-haemolytic Streptococci | Other beta haemolytic Streptococcus | beta Haemolytic Strep, group G |
| Beta-haemolytic Streptococci | Other beta haemolytic Streptococcus | beta Haemolytic Strep, not groups ABCDFG |
| Streptococcus pneumoniae | Streptococcus pneumoniae | Streptococcus pneumoniae |
| Other streptococcus spp. | S. anginosus group | Streptococcus anginosus |
| Other streptococcus spp. | S. anginosus group | Streptococcus constellatus |
| Other streptococcus spp. | S. anginosus group | Streptococcus intermedius |
| Other streptococcus spp. | Strep bovis group | Streptococcus bovis group |
| Other streptococcus spp. | Strep bovis group | Streptococcus equinus |
| Other streptococcus spp. | Strep bovis group | Streptococcus gallolyticus |
| Other streptococcus spp. | Strep bovis group | Streptococcus infantarius |
| Other streptococcus spp. | Strep bovis group | Streptococcus lutetiensis |
| Other streptococcus spp. | Nutritionally variant streptococci | Abiotrophia spp. |
| Other streptococcus spp. | Nutritionally variant streptococci | Granulicatella spp. |
| Other streptococcus spp. | Other streptococcus spp. | Streptococcus acidominimus |
| Other streptococcus spp. | Other streptococcus spp. | Streptococcus cristatus |
| Other streptococcus spp. | Other streptococcus spp. | Streptococcus gordonii |
| Other streptococcus spp. | Other streptococcus spp. | Streptococcus mitis |
| Other streptococcus spp. | Other streptococcus spp. | Streptococcus mutans |
| Other streptococcus spp. | Other streptococcus spp. | Streptococcus oralis |

| Other strentococcus snn | Streptococcus parasanguis |
|---|---|
| | Streptococcus pasteurianus |
| | Streptococcus salivarius |
| | Streptococcus sanguinis |
| · | |
| | Streptococcus sanguinus |
| | Streptococcus spp. |
| | Streptococcus uberis |
| | Streptococcus vestibularis |
| | Viridans Streptococcus |
| · | Enterococcus faecalis |
| - | Enterococcus faecium |
| · | Enterococcus spp. |
| | Escherichia coli |
| | Salmonella spp. |
| * * | Klebsiella aerogenes |
| * * | Klebsiella oxytoca |
| * * | Klebsiella ozaenae |
| | Klebsiella pneumoniae |
| | Klebsiella rhinoscleromatis |
| Klebsiella spp. | Klebsiella spp. |
| Other Enterobacterales | Citrobacter braakii |
| Other Enterobacterales | Citrobacter diversus |
| Other Enterobacterales | Citrobacter freundii |
| Other Enterobacterales | Citrobacter koseri |
| Other Enterobacterales | Citrobacter spp. |
| Other Enterobacterales | Citrobacter youngae |
| Other Enterobacterales | Enterobacter aerogenes |
| Other Enterobacterales | Enterobacter agglomerans |
| Other Enterobacterales | Enterobacter amnigenus |
| Other Enterobacterales | Enterobacter asburiae |
| Other Enterobacterales | Enterobacter cloacae |
| Other Enterobacterales | Enterobacter gergoviae |
| Other Enterobacterales | Enterobacter intermedius |
| Other Enterobacterales | Enterobacter sakazakii |
| Other Enterobacterales | Enterobacter spp. |
| Other Enterobacterales | Escherichia spp. |
| Other Enterobacterales | Hafnia alvei |
| Other Enterobacterales | Hafnia spp. |
| Other Enterobacterales | Kluyvera sp. |
| Other Enterobacterales | Morganella morganii |
| Other Enterobacterales | Morganella spp. |
| Other Enterobacterales | Pantoea agglomerans |
| | Pantoea spp. |
| | Proteus mirabilis |
| Other Enterobacterales | I TOLEUS ITIITUDIIIS |
| Other Enterobacterales Other Enterobacterales | Proteus spp. |
| | Other Enterobacterales |

| Other Enterobacterales | Other Enterobacterales | Providencia alcalifaciens |
|---|---|---|
| Other Enterobacterales | Other Enterobacterales | Providencia rettgeri |
| Other Enterobacterales | Other Enterobacterales | Providencia spp. |
| Other Enterobacterales | Other Enterobacterales | Providencia stuartii |
| Other Enteropacterales | Other Enteropacterales | Raoultella (Klebsiella) |
| Other Enterobacterales | Other Enterobacterales | ornithinolytica |
| Other Enterobacterales | Other Enterobacterales | Raoultella (Klebsiella) planticola |
| Other Enterobacterales | Other Enterobacterales | Raoultella (Klebsiella) terrigena |
| Other Enterobacterales | Other Enterobacterales | Serratia ficaria |
| Other Enterobacterales | Other Enterobacterales | Serratia liquefaciens |
| Other Enterobacterales | Other Enterobacterales | Serratia marcescens |
| Other Enterobacterales | Other Enterobacterales | Serratia odorifera |
| Other Enterobacterales | Other Enterobacterales | Serratia proteamaculans |
| Other Enterobacterales | Other Enterobacterales | Serratia rubidaea |
| Other Enterobacterales | Other Enterobacterales | Serratia spp. |
| Pseudomonas spp. | Pseudomonas aeruginosa | Pseudomonas aeruginosa |
| Pseudomonas spp. | Other <i>pseudomonas</i> spp. | Pseudomonas huttiensis |
| Pseudomonas spp. | Other <i>pseudomonas</i> spp. | Pseudomonas luteola |
| Pseudomonas spp. | Other <i>pseudomonas</i> spp. | Pseudomonas mallei |
| Pseudomonas spp. | Other <i>pseudomonas</i> spp. | Pseudomonas mendocina |
| Pseudomonas spp. | Other <i>pseudomonas</i> spp. | Pseudomonas oryzihabitans |
| Pseudomonas spp. | Other <i>pseudomonas</i> spp. | Pseudomonas pseudoalcaligenes |
| Pseudomonas spp. | Other <i>pseudomonas</i> spp. | Pseudomonas putida |
| Pseudomonas spp. | Other <i>pseudomonas</i> spp. | Pseudomonas spp. |
| Pseudomonas spp. | Other <i>pseudomonas</i> spp. | Pseudomonas stutzeri |
| Stenotrophomonas maltophilia | Stenotrophomonas maltophilia | Stenotrophomonas maltophilia |
| Acinetobacter spp. | Acinetobacter baumannii | Acinetobacter baumannii |
| Acinetobacter spp. | Other Acinetobacter spp. | Acinetobacter anitratus |
| Acinetobacter spp. | Other Acinetobacter spp. | Acinetobacter haemolyticus |
| Acinetobacter spp. | Other Acinetobacter spp. | Acinetobacter junii |
| Acinetobacter spp. | Other Acinetobacter spp. | Acinetobacter lwoffii |
| Acinetobacter spp. | Other Acinetobacter spp. | Acinetobacter radioresistens |
| Acinetobacter spp. | Other Acinetobacter spp. | Acinetobacter spp. |
| Anaerobic organism | Bacteroides spp. | Bacteroides spp. |
| Anaerobic organism | Clostridium spp. | Clostridium bifermentans |
| Anaerobic organism | Clostridium spp. | Clostridium botulinum |
| Anaerobic organism | Clostridium spp. | Clostridium butyricum |
| Anaerobic organism | Clostridium spp. | Clostridium cadaveris |
| Anaerobic organism | Clostridium spp. | Clostridium chauvei |
| Anaerobic organism | Clostridium spp. | Clostridium spp. |
| Anaerobic organism | Fusobacterium spp. | Fusobacterium necrophorum |
| Anaerobic organism | Fusobacterium spp. | Fusobacterium nucleatum |
| Anaerobic organism | Fusobacterium spp. | Fusobacterium spp. |
| Anaerobic organism | Porphyromonas spp. | Porphyromonas asacchrolytica |
| Anaerobic organism | Porphyromonas spp. | Porphyromonas gingivalis |
| Anaerobic organism | Porphyromonas spp. | Porphyromonas spp. |

| Anaerobic organism | Prevotella spp. | Prevotella spp. |
|---|---|---|
| Anaerobic organism | Anaerococcus spp. | Anaerococcus prevotii |
| Other bacteria | Actinomyces spp. | Actinomyces spp. |
| Other bacteria | Aerococcus spp. | Aerococcus spp. |
| Other bacteria | Aerococcus spp. | Aerococcus viridans |
| Other bacteria | Aeromonas spp. | Aeromonas caviae |
| Other bacteria | Aeromonas spp. | Aeromonas hydrophila |
| Other bacteria | Aeromonas spp. | Aeromonas sobria |
| Other bacteria | Aeromonas spp. | Aeromonas spp. |
| Other bacteria | | Aggregatibacter (Actinobacillus) |
| | Aggregatibacter spp. | actinomycetemcomitans |
| Other bacteria | Aggragatibastar.com | Aggregatibacter (Haemophilus) |
| Other bacteria | Aggregatibacter spp. | aphrophilus Aggregatibacter aphrophilus |
| Other bacteria | Aggregatibacter spp. | (Haemophilus paraphrophilus) |
| Other bacteria | Alcaligenes spp. | Alcaligenes dentrificans |
| Other bacteria | Alcaligenes spp. | Alcaligenes faecalis |
| Other bacteria | Alcaligenes spp. | Alcaligenes spp. |
| Other bacteria | Burkholderia spp. | Burkholderia cenocepacia |
| Other bacteria | Burkholderia spp. | Burkholderia cepacia |
| Other bacteria | Burkholderia spp. | Burkholderia cepacia complex |
| Other bacteria | Burkholderia spp. | Burkholderia gladioli |
| Other bacteria | Burkholderia spp. | Burkholderia multivorans |
| Other bacteria | Burkholderia spp. | Burkholderia spp. |
| Other bacteria | Burkholderia spp. | Burkholderia stabilis |
| Other bacteria | Burkholderia spp. | Burkholderia vietnamiensis |
| Other bacteria | Campylobacter spp. | Campylobacter fetus |
| Other bacteria | Campylobacter spp. | Campylobacter jejuni |
| Other bacteria | Campylobacter spp. | Campylobacter spp. |
| Other bacteria | Cardiobacterium spp. | Cardiobacterium hominis |
| Other bacteria | Cardiobacterium spp. | Cardiobacterium spp. |
| Other bacteria | Haemophilus spp. | Haemophilus influenzae |
| Other bacteria | Haemophilus spp. | Haemophilus spp. |
| Other bacteria | Listeria monocytogenes | Listeria monocytogenes |
| Other bacteria | Moraxella spp. | Moraxella catarrhalis |
| Other bacteria | Moraxella spp. | Moraxella lacunata |
| Other bacteria | Moraxella spp. | Moraxella osloensis |
| Other bacteria | Moraxella spp. | Moraxella spp. |
| Other bacteria | Neisseria gonorrhoeae | Neisseria gonorrhoeae |
| Other bacteria | Neisseria meningitidis | Neisseria meningitidis |
| Other bacteria | Pasteurella spp. | Pasteurella haemolytica |
| Other bacteria | Pasteurella spp. | Pasteurella multocida |
| Other bacteria | Pasteurella spp. | Pasteurella pneumotropica |
| Other bacteria | Pasteurella spp. | Pasteurella spp. |
| Other bacteria | Eikenella spp. | Eikenella corrodens |
| Other bacteria | Eikenella spp. | Eikenella spp. |
| Other bacteria | Any other | Rhodococcus spp. |

| Other bacteria | Any other | Actinobacillus spp. |
|---|---|---|
| Other bacteria | Any other | Arcanobacterium haemolyticum |
| Other bacteria | Any other | Aureobacterium spp. |
| Other bacteria | Any other | Capnocytophaga canimorsus |
| Other bacteria | Any other | Elizabethkingia meningoseptica |
| Other bacteria | Any other | Flavobacterium spp. |
| Other bacteria | Any other | Ralstonia mannitolilytica |
| Other bacteria | Any other | Ralstonia pickettii |
| Other bacteria | Any other | Ralstonia spp. |
| Other bacteria | Any other | Shewanella putrefaciens |
| Skin commensals other than | | |
| coagulase negative staph | Bacillus spp. | Bacillus spp. |
| Skin commensals other than | | |
| coagulase negative staph | Corynebacterium spp. | Corynebacterium spp. |
| Skin commensals other than | | |
| coagulase negative staph | Cutibacterium spp. | Cutibacterium acnes |
| Skin commensals other than | | |
| coagulase negative staph | Rhodococcus spp. | Rhodococcus equi |
| Skin commensals other than | | |
| coagulase negative staph | Rhodococcus spp. | Rhodococcus spp. |
| Skin commensals other than | | |
| coagulase negative staph | Dermabacter spp. | Dermbacter hominis |

## Appendix table 2. Antibiotic classes

| Antibiotic class | Antibiotic sub-class | Antibiotics |
|---|---|---|
| Penicillins | Natural penicillin | Phenoxymethylpenicillin |
| | | Benzylpenicillin |
| | Penicillinase-resistant penicillin | Flucloxacillin |
| | | Oxacillin |
| | | Methicillin |
| | Aminopenicillins (+/- beta- | Amoxicillin |
| | lactam inhibitor) | Ampicillin |
| | | Co-amoxiclav |
| | Mecillinam | Picmecillinam |
| | | Mecillinam |
| | Anti-pseudomonal penicillin | Piperacillin-tazobactam |
| | | Ticarcillin +/-beta-lactam |
| | Temocillin | Temocillin |
| Tetracyclines | First generation | Tetracycline |
| | | Oxytetracycline |
| | Second generation | Doxycycline |
| | | Lymecycline |
| | Glycylcyclines | Tigecycline |
| | Third generation tetracyclines | Eravacycline |
| | | Omadacycline |

| Cephalosporins | First generation | Cefalexin |
|---|---|---|
| cepnalosporms | That generation | Cefradine |
| | | Cefazolin |
| | Second generation | Cefuroxime |
| | Second generation | Cefaclor |
| | Third generation (+/- beta- | Ceración |
| | lactamase inhibitor) | Ceftriaxone |
| | lactariase initiation) | Cefotaxime |
| | | Ceftazidime |
| | Fourth generation (+/- beta- | Cefepime |
| | lactamase inhibitor) | · |
| | Fifth generation & siderophore | Ceftaroline |
| | | Ceftobiprole |
| | | Ceftolozane-tazobactam |
| | | Cefiderocol |
| Monobactam | | Aztreonam |
| Carbapenems (+/- beta | | Ertapenem |
| lactam inhibitors) | | Meropenem |
| | | Imipenem |
| Sulfonamides and | | Trimethroprim |
| Trimethoprim | | Co-trimoxazole |
| Macrolide | | Azithromycin |
| | | Erythromycin |
| | | Clarithromycin |
| Lincosamide | | Clindamycin |
| Aminoglycoside | | Gentamicin |
| | | Tobramycin |
| | | Amikacin |
| Quinolone/Fluroquinolone | | Nalidixic acid |
| | | Norfloxacin |
| | | Levofloxacin |
| | | Ciprofloxacin |
| | | Moxifloxacin |
| Glycopeptide | | Teicoplanin |
| | | Vancomycin |
| | | Dalbavancin |
| | Oxazolidinone | Linezolid |
| | Lipopeptide | Daptomycin |
| | Phosphonic acid | Fosfomycin |
| | Polymyxin | Colistin |
| | Imidazole | Metronidazole |
| | Nitrofuran | Nitrofurantoin |
| | Amphenicol | Chloramphenicol |
| | Rifamycin | Rifampicin |

- 1. Langford BJ, So M, Raybardhan S, et al. Antibiotic prescribing in patients with COVID-19: rapid review and meta-analysis. *Clin Microbiol Infect* 2021 doi: 10.1016/j.cmi.2020.12.018 [published Online First: 2021/01/09]
- 2. Langford BJ, So M, Raybardhan S, et al. Bacterial co-infection and secondary infection in patients with COVID-19: a living rapid review and meta-analysis. *Clin Microbiol Infect* 2020;26(12):1622-29. doi: 10.1016/j.cmi.2020.07.016 [published Online First: 2020/07/28]
- 3. Lansbury L, Lim B, Baskaran V, Lim WS. Co-infections in people with COVID-19: a systematic review and meta-analysis. *J Infect* 2020;81(2):266-75. doi: 10.1016/j.jinf.2020.05.046 [published Online First: 2020/05/31]
- 4. Rawson TM, Moore LSP, Zhu N, et al. Bacterial and Fungal Coinfection in Individuals With Coronavirus: A Rapid Review To Support COVID-19 Antimicrobial Prescribing. *Clin Infect Dis* 2020;71(9):2459-68. doi: 10.1093/cid/ciaa530 [published Online First: 2020/05/03]
- 5. Kaminsky LW, Dalessio S, Al-Shaikhly T, Al-Sadi R. Penicillin Allergy Label Increases Risk of Worse Clinical Outcomes in COVID-19. *J Allergy Clin Immunol Pract* 2021;9(10):3629-37 e2. doi: 10.1016/j.jaip.2021.06.054 [published Online First: 2021/07/23]
- 6. Sandoe JAT, Grozeva D, Albur M, et al. A retrospective propensity-score-matched cohort study of the impact of procalcitonin testing on antibiotic use in hospitalized patients during the first wave of COVID-19. *J Antimicrob Chemother* 2024;79(11):2792-800. doi: 10.1093/jac/dkae246
- 7. Benchimol EI, Smeeth L, Guttmann A, et al. The REporting of studies Conducted using Observational Routinely-collected health Data (RECORD) statement. *PLoS Med* 2015;12(10):e1001885. doi: 10.1371/journal.pmed.1001885 [published Online First: 2015/10/07]
- Docherty AB, Mulholland RH, Lone NI, et al. Changes in in-hospital mortality in the first wave of COVID-19: a multicentre prospective observational cohort study using the WHO Clinical Characterisation Protocol UK. *Lancet Respir Med* 2021;9(7):773-85. doi: 10.1016/S2213-2600(21)00175-2 [published Online First: 2021/05/18]
- 9. Suzuki E, Shinozaki T, Yamamoto E. Causal Diagrams: Pitfalls and Tips. *J Epidemiol* 2020;30(4):153-62. doi: 10.2188/jea.JE20190192 [published Online First: 20200201]
- 10. Cai L, Chen H, Wei Y, et al. Changing epidemiology, microbiology and mortality of bloodstream infections in patients with haematological malignancies before and during SARS-CoV-2 pandemic: a retrospective cohort study. BMJ Open 2023;13(12):e078510. doi: 10.1136/bmjopen-2023-078510 [published Online First: 20231230]
- 11. Santoro A, Franceschini E, Meschiari M, et al. Epidemiology and Risk Factors Associated With Mortality in Consecutive Patients With Bacterial Bloodstream Infection: Impact of MDR and XDR Bacteria. *Open Forum Infect Dis* 2020;7(11):ofaa461. doi: 10.1093/ofid/ofaa461 [published Online First: 20200930]
- 12. Gudiol C, Bodro M, Simonetti A, et al. Changing aetiology, clinical features, antimicrobial resistance, and outcomes of bloodstream infection in neutropenic cancer patients. *Clin Microbiol Infect* 2013;19(5):474-9. doi: 10.1111/j.1469-0691.2012.03879.x [published Online First: 20120424]
- 13. Magiorakos AP, Srinivasan A, Carey RB, et al. Multidrug-resistant, extensively drug-resistant and pandrug-resistant bacteria: an international expert proposal for interim standard definitions for acquired resistance. *Clin Microbiol Infect* 2012;18(3):268-81. doi: 10.1111/j.1469-0691.2011.03570.x [published Online First: 2011/07/29]
- 14. ATC/DDD Index WHO, 2024.

| 15. Bennet JE. Mandell, Douglas, and Bennett's Principles and Practice of Infectious Diseases. 9 ed: Elsevier 2015:251-496. |
|---|